CLINICAL TRIAL: NCT00681252
Title: Phase I/II Study of Multiple-Vaccine Therapy Using Epitope Peptide Restricted to HLA-A*0201 in Treating Patients With Refractory Gastric Cancer
Brief Title: Histocompatibility Leukocyte Antigen (HLA)-A*0201 Restricted Peptide Vaccine Therapy in Patients With Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tokyo University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Naohida Yamashita, MD/PhD, The Institute of Medical Science, The University of Tokyo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMS-MKA0201
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Gastric Cancer
Keywords: Peptide Vaccine; URLC10; VEGFR1; VEGFR2
MeSH Terms: conditions — Stomach Neoplasms | interventions — LY6K protein, human; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Biological: URLC10, VEGFR1 and VEGFR2

INTERVENTIONS:
Biological: URLC10, VEGFR1 and VEGFR2 — Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, the URLC10 peptide (1mg), VEGFR1 peptide (1mg) and VEGFR2 peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection in combination with S-1 chemotherapy.

SUMMARY:
The purpose of this study is to evaluate the safety and time to progression of HLA-A*0201 restricted epitope peptides URLC10, VEGFR1 and VEGFR2 emulsified with Montanide ISA 51.

DETAILED DESCRIPTION:
URLC10 has been identified as cancer specific molecules especially in non small cell lung cancer using genome-wide expression profile analysis by cDNA microarray technique. In a prior study, it has been shown that URLC10 is upregulated in human gastric tumors. VEGF receptor 1 and 2 are essential targets to tumor angiogenesis, and we identified that peptides derived from these receptors significantly induce the effective tumor specific CTL response in vitro and vivo. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of those peptides. Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, the URLC10-117 peptide (1mg), VEGFR1 peptide (1mg) and VEGFR2 peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection. The patients will also receive oral chemotherapy (S-1) simultaneously. Repeated cycles of vaccine will be administered until patients develop progressive disease or unacceptable toxicity, whichever occurs first. In the phase I study, we evaluate the safety and tolerability of these peptide vaccines. In the following phase II study, we evaluate the immunological and clinical response of this vaccine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent gastric cancer
* Resistant against conventional chemotherapy or difficult to continue the chemotherapy due to intolerable side effect(s)
* ECOG performance status 0-2
* Life expectancy > 3 months
* HLA-A*0201
* Laboratory values as follows 2000/mm3<WBC<15000/mm3 Platelet count>100000/mm3 Bilirubin < 3.0mg/dl Asparate transaminase < 150IU/L Alanine transaminase < 150IU/L Creatinine < 3.0mg/dl
* Able to receive oral TS-1 therapy
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy (woman of childbearing potential:Refusal or inability to use effective means of contraception)
* Breastfeeding
* Active or uncontrolled infection
* Unhealed external wound
* Concurrent treatment with steroids or immunosuppressing agent
* Prior chemotherapy, radiation therapy, and/or immunotherapy within 4 weeks
* Uncontrolled brain and/or intraspinal metastasis
* History of allergy to Tegaful, Gimeracil and/or Oteracil
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
safety (Phase I: toxicities as assessed by NCI CTCAE version 3) and efficacy (Phase II: Feasibility as evaluated by RECIST) | two months

SECONDARY OUTCOMES:
To evaluate immunological responses | two months

CONTACTS AND LOCATIONS:
Overall Officials: Naohide Yamashita, MD/PhD, Study Chair — Tokyo University
Locations (1):
- The Institutute of Medical Science, University of Tokyo, 4-6-1, Shirokanedai, Minato-ku, Tokyo, Japan

REFERENCES:
- [Background] Okabe H, Satoh S, Kato T, Kitahara O, Yanagawa R, Yamaoka Y, Tsunoda T, Furukawa Y, Nakamura Y. Genome-wide analysis of gene expression in human hepatocellular carcinomas using cDNA microarray: identification of genes involved in viral carcinogenesis and tumor progression. Cancer Res. 2001 Mar 1;61(5):2129-37. PMID 11280777
- [Background] Hasegawa S, Furukawa Y, Li M, Satoh S, Kato T, Watanabe T, Katagiri T, Tsunoda T, Yamaoka Y, Nakamura Y. Genome-wide analysis of gene expression in intestinal-type gastric cancers using a complementary DNA microarray representing 23,040 genes. Cancer Res. 2002 Dec 1;62(23):7012-7. PMID 12460921
- [Background] Takahashi M, Tsunoda T, Seiki M, Nakamura Y, Furukawa Y. Identification of membrane-type matrix metalloproteinase-1 as a target of the beta-catenin/Tcf4 complex in human colorectal cancers. Oncogene. 2002 Aug 29;21(38):5861-7. doi: 10.1038/sj.onc.1205755. PMID 12185585
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316